CLINICAL TRIAL: NCT05442515
Title: Phase 1/2 Dose Escalation Study of CD19/CD22 Bicistronic Chimeric Antigen Receptor (CAR) T Cells in Children and Young Adults With Recurrent or Refractory CD19/CD22-expressing B Cell Malignancies
Brief Title: CD19/CD22 Bicistronic Chimeric Antigen Receptor (CAR) T Cells in Children and Young Adults With Recurrent or Refractory CD19/CD22-expressing B Cell Malignancies
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10000324; 000324-C
Record Dates: First submitted 2022-07-01; First posted 2022-07-05 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07-25

CONDITIONS: B-NHL; B-Non Hodgkin Lymphoma; Acute Lymphocytic Leukemia; Acute Lymphoblastic Leukemia; B-precursor ALL; B-All; Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, B Cell; B-Cell Lymphoma; B-Cell Leukemia; Acute Lymphoid Leukemia
Keywords: Philadelphia chromosome + ALL; Lymphoma; CD-22 Expressing Tumor; CD-19 expressing tumor; Adoptive Immunotherapy; B-All; B-precursor ALL; Acute Lymphoblastic Leukemia; Acute Lymphocytic Leukemia; B-Non Hodgkin Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Lymphoma, Non-Hodgkin; Leukemia, B-Cell; Lymphoma, B-Cell; Philadelphia Chromosome; Lymphoma | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- 1/Phase I Dose Escalation-with standard LD - CLOSED (Experimental): CD19/CD22-CAR-transduced T cells at escalating dose + standard LD
  Interventions: Biological: CD19/CD22-CAR-transduced T cells; Drug: cyclophosphamide; Drug: fludarabine
- 1b/Phase 1 Dose Escalation - low disease burden (Experimental): CD19/CD22-CAR-transduced T cells
  Interventions: Biological: CD19/CD22-CAR-transduced T cells; Drug: cyclophosphamide; Drug: fludarabine
- 2/Phase I Dose Escalation- with intensified LD - CLOSED (Experimental): CD19/CD22-CAR-transduced T cells + standard LD
  Interventions: Biological: CD19/CD22-CAR-transduced T cells; Drug: cyclophosphamide; Drug: fludarabine
- 2b/Phase 1 Dose Escalation - high disease burden (Experimental): CD19/CD22-CAR-transduced T cells
  Interventions: Biological: CD19/CD22-CAR-transduced T cells; Drug: cyclophosphamide; Drug: fludarabine
- 3/Phase II Dose Expansion- with low disease burden (Experimental): CD19/CD22-CAR-transduced T cells at MTD/or highest dose administered with LD
  Interventions: Biological: CD19/CD22-CAR-transduced T cells; Drug: cyclophosphamide; Drug: fludarabine
- 4/Phase II Dose Expansion- with high disease burden (Experimental): CD19/CD22-CAR-transduced T cells at MTD/or highest dose administered with LD regimen #2
  Interventions: Biological: CD19/CD22-CAR-transduced T cells; Drug: cyclophosphamide; Drug: fludarabine
- A/Pre-treatment (No Intervention): All participants enrolled on the study prior to treatment initiation.

INTERVENTIONS:
Biological: CD19/CD22-CAR-transduced T cells — CD19/CD22-CAR-transduced T cells on D0 after lymphodepleting preparative regimen
  Arms: 1/Phase I Dose Escalation-with standard LD - CLOSED; 1b/Phase 1 Dose Escalation - low disease burden; 2/Phase I Dose Escalation- with intensified LD - CLOSED; 2b/Phase 1 Dose Escalation - high disease burden; 3/Phase II Dose Expansion- with low disease burden; 4/Phase II Dose Expansion- with high disease burden
Drug: cyclophosphamide — Cyclophosphamide will be diluted in an appropriate solution and infused over one hour. The dose will be based on the patient s body weight, at 900 mg/m2/dose after fludarabine infusion.
  Arms: 1/Phase I Dose Escalation-with standard LD - CLOSED; 1b/Phase 1 Dose Escalation - low disease burden; 2/Phase I Dose Escalation- with intensified LD - CLOSED; 2b/Phase 1 Dose Escalation - high disease burden; 3/Phase II Dose Expansion- with low disease burden; 4/Phase II Dose Expansion- with high disease burden
Drug: fludarabine — Fludarabine is administered as an IV infusion in an appropriate solution over 30 minutes. To prevent undue toxicity the dose will be based on BSA (25 mg/m2/dose).
  Arms: 1/Phase I Dose Escalation-with standard LD - CLOSED; 1b/Phase 1 Dose Escalation - low disease burden; 2/Phase I Dose Escalation- with intensified LD - CLOSED; 2b/Phase 1 Dose Escalation - high disease burden; 3/Phase II Dose Expansion- with low disease burden; 4/Phase II Dose Expansion- with high disease burden

SUMMARY:
Background:

Acute lymphoblastic leukemia (ALL) is the most common cancer in children. About 90% of children and young adults who are treated for ALL can now be cured. But if the disease comes back, the survival rate drops to less than 50%. Better treatments are needed for ALL relapses.

Objective:

To test chimeric antigen receptor (CAR) therapy. CARs are genetically modified cells created from each patient s own blood cells. his trial will use a new type of CAR T-cell that is targeting both CD19 and CD22 at the same time. CD19 and CD22 are proteins found on the surface of most types of ALL.

Eligibility:

People aged 3 to 39 with ALL or related B-cell lymphoma that has not been cured by standard therapy.

Design:

Participants will be screened. This will include:

Physical exam

Blood and urine tests

Tests of their lung and heart function

Imaging scans

Bone marrow biopsy. A large needle will be inserted into the body to draw some tissues from the interior of a bone.

Lumbar puncture. A needle will be inserted into the lower back to draw fluid from the area around the spinal cord.

Participants will undergo apheresis. Their blood will circulate through a machine that separates blood into different parts. The portion containing T cells will be collected; the remaining cells and fluids will be returned to the body. The T cells will be changed in a laboratory to make them better at fighting cancer cells.

Participants will receive chemotherapy starting 4 or 5 days before the CAR treatment.

Participants will be admitted to the hospital. Their own modified T cells will be returned to their body.

Participants will visit the clinic 2 times a week for 28 days after treatment. Follow-up will continue for 15 years....

DETAILED DESCRIPTION:
Background:

* Despite improvements in therapy, acute lymphoblastic leukemia (ALL) contributes to significant morbidity and mortality for children and young adults with cancer. CD19-CAR and CD22-CAR therapy have proven highly effective in inducing remission in patients with relapsed/refractory disease.
* Immune escape has been observed by several groups following CD19-CAR and CD22- CAR therapy for B-ALL. Investigation of this phenomenon reveals a complex biology responsible for loss or downregulation of CD19 and/or CD22 expression observed in these cases.
* The challenges encountered with currently available CD19- and CD22-directed CAR T cells in B-ALL demonstrates the need for combinatorial treatment strategies simultaneously targeting two antigens, such as CD19 and CD22, to enhance the long-term effectiveness of CARs.
* We have previously treated patients with B-ALL on a phase 1/2 clinical trial using a bivalent CD19/22 CAR T-cell as a first combinatorial treatment strategy. This CAR T-cell construct is well-tolerated and has yielded responses however there has been limited CAR T cell expansion and persistence. Additionally, the previously tested CD19/CD22 bivalent CAR T-cell construct is limited in its ability to target CD22.
* This new CD19/22 targeted construct being tested in this clinical trial has improved dual targeting capability based on preclinical data/evaluation.

Objectives:

* Phase I: Assess the safety of administering escalating doses of autologous CD19/CD22- CAR engineered T cells in children and young adults with B cell ALL (stratified by disease burden) or lymphoma following a cyclophosphamide/fludarabine conditioning regimen.
* Phase II: Determine the efficacy of CD19/CD22 therapy in participants stratified by disease burden.

Eligibility:

-Participants between >= 3 years and <= 39 years of age, with CD19+/CD22+ B cell ALL or lymphoma who have relapsed or have refractory disease after at least one standard chemotherapy regimen and one salvage regimen, with no alternative curative options.

Design:

* Phase I, 3 + 3 dose escalation design across 3 cohorts (B-ALL/B-cell lymphoblastic lymphoma: A: low-disease burden (<25 % marrow blasts without extramedullary disease) vs. B: high-disease burden (>= 25 % marrow blasts or with EMD): C: B-cell non-Hodgkin lymphoma using the following dose levels: -2: 1 x 10^5 transduced T cells/kg (+/- 20%); -1: 3 x 10^5 transduced T cells/kg (+/- 20%); 1: 1 x 10^6 transduced T cells/kg (+/- 20%); and 2: 3x 10^6 transduced T cells/kg (+/- 20%). Cohorts will enroll concurrently.
* Participants will be treated based on disease burden and will receive 1 of 2 lymphodepleting preparative regimens:

  * Lymphodepleting preparative regimen # 1: Fludarabine (30 mg/m^2/d x 3 on Days -4, -3, -2) and cyclophosphamide (900 mg/m^2/d x 1 on Day -2) followed by infusion of CD19/CD22-CAR T-cells on D0.
  * Lymphodepleting preparative regimen #2: Fludarabine (30 mg/m2/d x 4 on Days -5, -4, -3, -2) and cyclophosphamide (600 mg/m2/d x 2 on Days -3, -2) followed by infusion of CD19/CD22-CAR T-cells on D0.
  * Determination for use of LD regimen #1 versus #2 will be based on pre-treatment absolute lymphocyte count, pre-existing cytopenias, receipt of prior CAR T-cell therapy, high disease burden and assessment of infection risk.
* Participants will be evaluated sequentially for toxicity, antitumor effects, CAR expansion and persistence, and other biologic correlatives.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Diagnosis

  * Participant must:

    * Have pathology confirmed B cell ALL (not isolated to the testis or CNS), CML with ALL transformation, or high-grade lymphoma (e.g., Burkitt's lymphoma, B-lymphoblastic lymphoma, diffuse large B-cell lymphoma, inclusive of low-grade lymphoma that has transformed to high grade disease); and
    * Have relapsed or been refractory after at least one standard chemotherapy regimen and at least one salvage treatment. Participants with Philadelphia chromosome + ALL must have failed prior tyrosine kinase inhibitor; and
    * Be ineligible for allogeneic stem cell transplant (SCT), have refused SCT, or have recurred after SCT; and
    * Have no evidence of graft-versus- host disease (GVHD) and have been without immunosuppressive agents for at least 30 days prior to apheresis, if undergone prior allogeneic SCT; and
    * Be unable to access (in a timely manner), ineligible for, or have relapsed/failed after or not responded to a commercially available CD19 CAR T-cell construct; and
  * Have evidence of at least minimal residual disease or PET-avid disease (lymphoma) at the time of enrollment.
* CD22/CD19 expression

  * CD19 must be detected on >15% of the malignant cells by immunohistochemistry or > 80% by flow cytometry.
  * CD22 positivity must be confirmed.
* Age >= 3 years of age and <=39 years of age at time of enrollment.
* Clinical Performance status: Participants >= 16 years of age: Karnofsky >= 50%; Participants < 16 years of age: Lansky scale >= 50%.
* Participants must have adequate organ and marrow function as defined below:

  * leukocytes >= 750/mcL*
  * platelets >= 50,000/mcL*
  * total bilirubin <=2 X ULN (except in the case of participants with documented Gilbert's disease > 3x ULN)
  * AST(SGOT)/ALT(SGPT) <=10 X institutional upper limit of normal
  * creatinine <= the maximum for age listed in the table below OR
  * measured creatinine clearance >=60 mL/min/1.73 m^2 for participants with creatinine levels above the max listed below per age.

    * Age (Years) <= 5 / Maximum Serum Creatinine (mg/dL) <= 0.8
    * Age (Years) 6 to <= 10 / Maximum Serum Creatinine (mg/dL) <= 1.0
    * Age (Years) >10 / Maximum Serum Creatinine (mg/dL) <= 1.2

      * a participant will not be excluded because of pancytopenia >= Grade 3 if it is due to underlying bone marrow involvement by leukemia
* Central nervous system (CNS) Status
* Participants with leukemia with CNS 1 and 2 disease are eligible in the absence of exclusion criteria
* Participants of child-bearing or child-fathering potential must be willing to practice effective birth control from the time of enrollment until 12 months following completion of study treatment for women and for 4 months following completion of study treatment for men.
* Participants who are breastfeeding or plan to breastfeed must agree to discontinue/postpone breastfeeding while on study therapy and until 1 month after the administration of CAR.
* Cardiac function: Left ventricular ejection fraction >= 45% or fractional shortening >=28%
* Pulmonary Function

  * Baseline oxygen saturation >92% on room air at rest
* Ability of participant or Legally Authorized Representative (LAR) to understand and the willingness to sign a written informed consent document.
* Ability and willingness of participant or Legally Authorized Representative (LAR) to co- enroll on 15-C-0028: Follow-up Evaluation for Gene-Therapy Related Delayed Adverse Events after Participation in Pediatric Oncology Branch Clinical Trials.

EXCLUSION CRITERIA:

Participants meeting any of the following criteria are not eligible for participation in the study:

* Participants with CNS3 disease, progressing neurologic signs* of CNS disease, radiologically detected active CNS lymphoma (*resolving manifestation or persistent and/or irreversible findings from prior CNS involvement (e.g., blindness) is not exclusionary)
* Hyperleukocytosis (>= 50,000 blasts/microL)
* Positive serum or urine beta-HCG pregnancy test performed at screening.
* Participants will be excluded based on prior therapy if they fail to meet following washout criteria:

  * Therapy: Systemic Chemotherapy, anti-neoplastic agents, antibody- based therapies
  * Washout*: >=2 weeks
  * Exceptions: 6 weeks for clofarabine or nitrosoureas; No washout for prior intrathecal chemotherapy, steroid therapy, hydroxyurea (no dose increases within prior 2 weeks) or ALL maintenance-type chemotherapy (vincristine, 6-mercaptopurine, oral methotrexate, or a tyrosine kinase inhibitor for participants with Ph+ ALL) provided there is recovery from any acute toxic effects
  * Therapy: Radiation
  * Washout*: >=3 weeks
  * Exceptions: No time restriction with radiation therapy if the volume of bone marrow treated is less than 10% and the participant has measurable/evaluable disease outside the radiation window
  * Therapy: Allogeneic Stem Cell Transplant
  * Washout*: >= 100 days since SCT; >= 30 days since completion of immunosuppression; >= 6 weeks since donor lymphocyte infusion (DLI)
  * Exceptions: Cannot have evidence of active graft-versus-host disease (GVHD)
  * Therapy: CAR T-Cell Therapy or other Adoptive Cell Therapy
  * Washout*: > 30 days post infusion

    * Washout: Time between therapy and apheresis
* Positive HIV antibodies consistent with active HIV.
* Positive hepatitis C antibodies or positive Hepatitis B surface antigen (HbsAG) indicative of current/active HCV/HBV.
* Active second malignancy other than in situ carcinoma of the cervix, unless the tumor was treated with curative intent at least two years previously and participant is in remission.
* History of severe, immediate hypersensitivity reaction attributed to compounds of similar chemical or biologic composition to any agents used in study or in the manufacturing of the cells.
* Uncontrolled, symptomatic, intercurrent illness or social situations that would limit compliance with study requirements or in the opinion of the PI would pose an unacceptable risk to the participant.

Ages: 3 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 126 (Estimated)
Dates: Start 2022-12-28 (Actual); Primary Completion 2027-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy | Monthly until 3 months post CAR T infusion and then at 6 months and every 6 months after that, for 2 years post-infusion for each participant, up to 2 years after the entry date of the last participant.
  Determine the efficacy of CD19/CD22 therapy in participants stratified by disease burden.
Safety | 30 days post CAR T infusion
  Assess the safety of administering escalating doses of autologous CD19/CD22-CAR engineered T cells in children and young adult with B cell ALL (stratified by disease burden) or lymphoma following a cyclophosphamide/fludarabine LD.

SECONDARY OUTCOMES:
Feasibility | Up to two years after the last participant has entered.
  Determine the feasibility of producing CD19/CD22-CAR T cells meeting the established release criteria.
Adverse Events | 30 days post CAR T infusion
  Phase II: Assess the safety of CD19/CD22 therapy in participants based on underlying disease burden.
Persistence and expansion | Up to two years after the last participant has entered.
  Evaluate persistence and expansion of C19/CD22-CAR T cells in children and young adults with CD19+CD22+ B-ALL or lymphoma
Progression free survival (PFS) and Overall survival (OS) | Up to two years after the last participant has entered.
  Evaluate PFS and OS in participants, separately by phase II cohort
Overall response rate | Monthly until 3 months post infusion and then at 6 months and every 6 months after that, for 2 years post-infusion for each participant, for up to two years from the entry date of the last participant
  Phase I: Evaluate the ability of CD19/CD22-CAR T cells to mediate clinical activity in children and young adults with CD19+CD22+ B cell ALL or lymphoma.
Assess response and toxicity (CRS grade) | Up to two years after last participant has entered
  Assess overall response rate and CRS grades (toxicity) in participants who received subsequent infusion

CONTACTS AND LOCATIONS:
Overall Officials: Nirali N Shah, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000324-C.html